CLINICAL TRIAL: NCT04968015
Title: A Phase II Randomized Study to Assess the Efficacy on Outcome of Venetoclax Combined With Cytarabine Versus Idarubicin Combined With Cytarabine Administered as Post-remission Therapy to Elderly Patients With Acute Myeloid Leukemia in First Remission
Brief Title: Venetoclax + Cytarabine Versus Idarubicin + Cytarabine : Efficacity Assessment as Post-remission Therapy to Elderly Patients With Acute Myeloid Leukemia in First Remission
Acronym: LAMSA2020
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAMSA2020
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Phase II open label controlled study. Subjects will be randomized 1:1 to receive Venetoclax or Idarubicin associated to Cytarabine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VEN-CYTA (Experimental): Venetoclax 600mg/day, Per Os (PO), D1 to D14 / 28 days cycle Cytarabine 50 mg/m2/12h Subcutaneous (SC), D1 to D5 / 28 days cycle
  Interventions: Drug: Cytarabine-Venetoclax Association
- IDA-CYTA (Active Comparator): Idarubicin 8mg/m2, Intravenous (IV), at D1 / 28 days cycle Cytarabine 50 mg/m2/12h, SC, D1 to D5 / 28 days cycle
  Interventions: Drug: Cytarabine-Idarubicin Association

INTERVENTIONS:
Drug: Cytarabine-Venetoclax Association — Consolidation treatment with cytarabine + venetoclax
  Arms: VEN-CYTA
Drug: Cytarabine-Idarubicin Association — Consolidation treatment with cytarabine + idarubicin
  Arms: IDA-CYTA

SUMMARY:
For the FILO group, the standard of care for induction chemotherapy of elderly fit patients with AML is represented by the combination of Cytarabine, Idarubicin and Lomustine. The superiority of this combination was confirmed in a larger prospective study the LAMSA-2007. This induction treatment, followed by six courses of consolidation (Idarubicin and Cytarabine) followed then by a period of 6-month maintenance therapy, allows up to 80 % of remission, and a RFS of 46 % at 2 years.

The aim of the study is to assess the efficacy on outcome of Venetoclax combined with Cytarabine versus Idarubicin combined with Cytarabine administered as post-remission therapy to elderly patients with acute myeloid leukemia in first complete remission (CR) following induction chemotherapy.

DETAILED DESCRIPTION:
Acute myeloid leukemia is characterized by the clonal expansion of myeloid blasts in the bone marrow, peripheral blood and extramedullary tissues which disrupts normal hematopoiesis.

It is the most common form of acute leukemia in adults with an estimated 19,950 new cases and 10,430 deaths in 2016 in the United States. The prevalence is approximately 36,000 in the US alone. The median age of diagnosis is 67 years, with 55 % of the patients diagnosed at 65 years or older, and approximately a third of them are diagnosed over the age of 75.

Due to a higher frequency of poor prognosis factors such as adverse cytogenetics, previous history of myelodysplastic syndrome (MDS) or therapy-related AML (t-AML), the prognosis of elderly AML remains dismal in patients > 60 years.

The complete remission rate achieved after induction chemotherapy is lower than in young adults, and the remission duration is seldom longer than a year. Consequently, the overall survival of these patients rarely excesses 10-15 % beyond 5 years from diagnosis. For this group of patients, improving the efficacy of post induction chemotherapy and preventing relapse, without increasing the treatment-related mortality, remain a challenge.

For the FILO group, the standard of care for induction chemotherapy of elderly fit patients with AML is represented by the combination of Cytarabine, Idarubicin and Lomustine (ICL: Idarubicin 8 mg per square meter per day, IV on days 1-5, Cytarabine 100 mg per square meter per day on days 1-7 IV continuously, Lomustine 200 mg per square meter orally at day 1). This induction treatment, followed by six courses of consolidation, consisting of reduced doses of Idarubicin 8 mg per square meter per day IV on day 1 and Cytarabine 50 mg per square meter/12h/d subcutaneously on days 1-5 followed then by a period of 6-month maintenance therapy, allows up to 80 % of remission, an improvement in 2-year Event Free Survival from 26 % to 41 %, and a 2 year relapse free survival improvement from of 33 % to 46 % for patients without unfavorable cytogenetics.

Venetoclax is a potent, selective and orally bioavailable small molecule inhibitor of BCL-2 (B-cell lymphoma 2), an anti-apoptotic protein which overexpression is associated with tumor initiation, disease progression, and drug resistance, and is thus a compelling target for anti-tumor therapy. Phse I/II studies have assessed venetoclax as single agent or in combination with low dose Cytarabine (LDAC) in upfront treatment of AML patients aged ≥ 65 years old and not eligible for standard Cytarabine and anthracycline-based induction therapy with encouraging results. The aim of the study is to assess the efficacy on outcome of Venetoclax combined with Cytarabine versus Idarubicin combined with Cytarabine administered as post-remission therapy to elderly patients with acute myeloid leukemia in first complete remission (CR) following induction chemotherapy.

Subjects will be randomized 1:1 to receive Venetoclax or Idarubicin associated to Cytarabine for 6 cycles x 28 days. Patients will be followed until progression or death or until the end of study defined by the number of relapse-free survival (RFS) events and last patient treatment period.

ELIGIBILITY:
Inclusion Criteria :

* ≥ 60 years of age.
* AML de novo according to the WHO 2016 classification
* AML with favorable or intermediate cytogenetics according to ELN 2017
* Subjects should be eligible for intensive chemotherapy by Idarubicin, Cytarabine, and Lomustine (standard induction for FILO)
* SORROR < 3 (for the protocol, calculation of Sorror excludes a history of cancer) (appendix 2)
* AML secondary to MDS or chemotherapy are eligible, unless adverse cytogenetics
* Eastern Cooperative Oncology Group (ECOG) < 3 (appendix 1)
* Adequate baseline organ function defined by the criteria below:

  * Adequate renal function as demonstrated by a creatinine clearance ≥ 50 mL/min; calculated by the Cockcroft Gault formula or measured by 24-hours urine collection
  * Aspartate aminotransferase (AST) ≤ 3.0 × upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) ≤ 3.0 × ULN
  * Bilirubin ≤ 1.5 × ULN
* Adequate cardiac function with Left Ventricular Ejection Fraction (LVEF) ≥ 50 %
* Absence of any psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule
* Females must be menopausal to be pre-enrolled
* Patients must be affiliated to the French Social Security (health insurance)
* Signed written informed consent for the study

Exclusion Criteria:

* Diagnosis of Acute Promyelocytic Leukemia (APL)
* AML with adverse cytogenetics according to ELN 2017
* AML with BCR-ABL1 translocation
* Subject with an antecedent of myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocytosis, polycythemia vera, or chronic myelogenous leukemia (CML) with or without BCR-ABL1 translocation
* Clinical symptoms suggesting active central nervous system leukemia, or presence of isolated extramedullary leukemia
* Previous exposure of anthracycline ≥ 550 mg/m² (Daunorubicin equivalence)
* Previous AML treatment other than Hydroxyurea
* Treatment with an investigational drug within 30 days or 5 half-life whichever is longer, preceding the initiation study and/or previous treatment with Venetoclax
* History of another malignancy within the past 3 years except basal cell carcinoma of the skin or cervix in situ carcinoma
* Any serious medical condition, laboratory abnormalities or psychiatric illness that would place the participant at an unacceptable risk or prevent them from giving informed consent or precluding the administration of protocol treatments
* Other comorbidity that the physician judges to be incompatible with conventional intensive chemotherapy which must be reviewed and approved by the study medical monitor before study enrolment
* Subject with known HIV infection (due to potential drug-drug interactions between antiretroviral medications and Venetoclax). HIV testing will be performed at Screening. Subject known to be positive for hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status with undetectable Polymerase Chain Reaction (PCR) viral load on antivirals (non-exclusionary medications) are not excluded.

Randomization criteria:

1. Subjects must have been registered at diagnosis
2. Subjects must have received intensive induction by Idarubicin, Cytarabine and Lomustine
3. Patients in Complete Response / Complete Response with incomplete hematologic recovery (CR/CRi) post induction according to ELN 2017 criteria
4. Randomization should be performed no more than D+60 after induction
5. ECOG < 3 (appendix 1)
6. Adequate baseline organ function defined by the criteria below:

   * Adequate renal function as demonstrated by a creatinine clearance ≥ 50 mL/min; calculated by the Cockcroft Gault formula or measured by 24-hours urine collection
   * Aspartate aminotransferase (AST) ≤ 3.0 × ULN
   * Alanine aminotransferase (ALT) ≤ 3.0 × ULN
   * Bilirubin ≤ 1.5 × ULN
7. Adequate cardiac function with LVEF ≥ 50 %
8. Male subjects who are sexually active must agree, from study Day 1 through at least 180 days after the last dose of study drug, to practice protocol-specified methods of contraception
9. Female subjects must be postmenopausal defined as with no menses for 12 or more months without an alternative medical cause

Non randomization criteria

1. Patient in Partial Remission (PR) or failure following one induction course by Idarubicin, Cytarabine and Lomustine (according ELN 2017 criteria)
2. Uncontrolled infection
3. Subject with cardiovascular disability status as per New York Heart Association Class > 2. Class 2 is defined as cardiac disease in which subjects are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or angina pain. Class 3 is defined as cardiac disease in which subjects are comfortable at rest but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class 4 is defined as cardiac disease in which subjects have an inability to carry on any physical activity without discomfort, symptoms of heart failure at rest, and if any physical activity is undertaken then discomfort increases.
4. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration.
5. Any serious medical condition, laboratory abnormality, or psychiatric illness that would place the participant at an unacceptable risk or prevent them from giving informed consent.
6. Treatment with any of the following within 7 days prior to the first dose of study drug :

   * Strong or moderate CYP3A inducers
   * Steroid therapy for anti-neoplastic intent
7. Subject having consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment.
8. Subject having chronic respiratory disease that requires continuous oxygen, or a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
9. Previous treatment with Venetoclax and/or current participation in any other research study with investigational products.
10. Known hypersensitivity to the study medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival (RFS) | from randomization to last follow-up (up to 5 years)
  RFS measured from the date of achievement of a remission until the date of relapse or death from any cause

SECONDARY OUTCOMES:
Overall survival at 2 years | from date of randomization to 2 years after last administration of experimental treatment
  time from date of randomization to date of death

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud PIGNEUX, Pr, Principal Investigator — FILO (French Innovative Leukemia Organization); Yosr HICHERI, Principal Investigator — FILO (French Innovative Leukemia Organization)
Locations (26):
- France (26):
  - ANGERS - CHU - Maladies du sang, Angers
  - ANNECY - Centre Hospitalier Annecy-Genevois, Annecy
  - AVIGNON - Centre Hospitalier, Avignon
  - BAYONNE - CH de la Côte Basque - Hématologie, Bayonne
  - BESANCON - Hôpital Jean Minjoz - Hématologie, Besançon
  - BEZIERS - Centre Hospitalier - Hématologie, Béziers
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - Grenoble - CHUGA - Hématologie Clinique, Grenoble
  - LYON-Centre Léon Bérard, Lyon
  - MARSEILLE - Institut Paoli-Calmettes, Marseille
  - METZ - CHR Metz-Thionville, Metz
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - MULHOUSE - Hôpital E. Muller - Hématologie, Mulhouse
  - NANTES - Hôpital Hôtel Dieu - Hématologie Clinique, Nantes
  - NIMES - CHU Caremeau, Nîmes
  - ORLEANS - CHR - Hématologie, Orléans
  - PERPIGNAN - CH St Jean - Hématologie Clinique, Perpignan
  - BORDEAUX - Hôpital Haut-Levêque, Pessac
  - POITIERS - Hôpital La Milétrie - Hématologie Clinique, Poitiers
  - REIMS - Hôpital Robert Debré - Hématologie Clinique, Reims
  - RENNES - Hôpital Pontchaillou - Hématologie, Rennes
  - ST ETIENNE - CHU et Institut De Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - NANCY - CHU de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided